CLINICAL TRIAL: NCT02856529
Title: Effects of Basic Infection Control Skills License on Knowledge and Practice of Health Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Madinah Saudi Board Community Medicine (Other Government)
Collaborators: Madinah directorate - Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBCMM001
Record Dates: First submitted 2016-06-18; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Infection Control Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): A BICSL certified trainer conduct the intervention. It includes hand on training session standardized in a scientific way. The participants trained on hand hygiene and use of PPE. Also, it includes meningitis and influenza vaccination as well as fit test to verify the correctly fitting of the respirator.
  Interventions: Other: Training
- Control (Active Comparator): A general session about the basic of infection control was conducted for this group. The lecture performed in the same way of the regular training fulfill.
  Interventions: Other: General session

INTERVENTIONS:
Other: Training — The Basic Infection Control Skills License program (BICSL) includes meningitis and influenza vaccination as well as fit test to verify the correctly fitting of the respirator. Also, the license program includes training on hand hygiene and the use of personal protective equipment (PPE). To get the license, each participants must get the vaccination and attend one to one training session with a program trainer 34.
  Arms: Intervention
Other: General session — A general session about the basic of infection control was conducted for this group. The lecture performed in the same way of the regular training fulfill.
  Arms: Control

SUMMARY:
Considering the importance of infection control practices, Madinah Public Health Department launched a new license program for healthcare workers, the Basic Infection Control Skills License program (BICSL). BICSL has been launched to train healthcare workers all over the region in a scientific standardized way.

To assess BICSL effectiveness, a non-randomized control study will be conducted in two of the general hospitals in Madinah. An electronic bilingual self-administrated valid and reliable questionnaire will be used to evaluate the workers knowledge and practices before and after three and six months of the intervention. The knowledge and practice answers were scored and the scores were categorized to facilitate the comparison. A BICSL certified trainer will be conducting the intervention, a one to one training session. A SPSS program will be used to analyze the data. Administrative and ethical approval was obtained from Madinah health authority. The participants will complete an electronic consent before they fill the questionnaire. Confidentiality and privacy as well as freedom to participate or not will be insured to all participants. This study will assess the license effectiveness in improve knowledge and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Working in the chosen hospitals.
2. Health care worker (Physician, nurse or technician) of any gender, age, or experience.

Exclusion Criteria:

1. Refuse to participate in the study.
2. Have BICSL certificate before the study implemented.
3. On leave during study period.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Self administered knowledge | 3 months
  will be measured by questionnaire
Self administered practice | 3 months
  will be measured by questionnaire

SECONDARY OUTCOMES:
Self administered knowledge | 3 months
  between different sexes and professions, it will be measured by questionnaire
Self administred practices | 3 months
  between different sexes and professions, it will be measured by questionnaire

IPD SHARING:
Plan to Share IPD: No